CLINICAL TRIAL: NCT06464406
Title: Effects of Virtual Reality on Cardiorespiratory Fitness Test Results
Brief Title: Virtual Reality During Exercise Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Andrew Moore, Assistant Professor, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2130870
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Virtual Reality
Keywords: virtual reality; cardiorespiratory fitness; anaerobic threshold; bicycle ergometer test

STUDY DESIGN:
Intervention Model Description: This study will use a repeated-measures crossover model in which each participant completes the two conditions of the maximal exercise test (Control and Virtual Reality) in a randomized, counterbalanced order.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to mask the participant or data collection personnel from the conditions because the Virtual Reality condition requires that the headset be worn. Metabolic data and resulting outcomes (i.e. VO2peak value) will be analyzed by independent research assistants who will be blinded to the condition under which the data were gathered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control condition completed first (Experimental): In this arm, the Control condition (traditional maximal cardiorespiratory exercise test) will be completed first, and the Virtual Reality condition (traditional maximal cardiorespiratory exercise test with the addition of virtual reality video) will be completed second.
  Interventions: Behavioral: Virtual Reality condition; Behavioral: Control condition
- Virtual Reality condition completed first (Experimental): In this arm, the Virtual Reality condition (traditional maximal cardiorespiratory exercise test with the addition of virtual reality video) will be completed first, and the Control condition (traditional maximal cardiorespiratory exercise test) will be completed second.
  Interventions: Behavioral: Virtual Reality condition; Behavioral: Control condition

INTERVENTIONS:
Behavioral: Virtual Reality condition — Participants will watch a video on a virtual reality headset during the completion of the maximal cardiorespiratory exercise test.
Behavioral: Control condition — Participants will complete the maximal cardiorespiratory exercise test under control conditions without video, music, or other distractions.

SUMMARY:
The goal of this clinical trial is to explore the effects of virtual reality use on maximal aerobic exercise test performance (aerobic capacity) in healthy adults. The main questions it aims to answer are:

* Does using a virtual reality program during a maximal aerobic exercise test lead to differences in VO2peak (maximal aerobic capacity)? and,
* Does using a virtual reality program during a maximal aerobic exercise test lead to differences in work rate at the ventilatory threshold?

Participants will complete a maximal aerobic exercise test two times (separated by 1 week of recovery) under the following conditions:

* normal testing conditions in a lab
* while viewing a virtual reality video

Researchers will compare the test results of both conditions to see if the use of a virtual reality program alters VO2peak or the ventilatory threshold.

DETAILED DESCRIPTION:
Virtual reality imparts a dissociative effect on users during exercise, such that the physical activity task is experienced as more enjoyable and pleasant, requires less exertion, and requires less physiological function for a given submaximal work rate.

This array of positive effects may be particularly advantageous during a maximal aerobic exercise test, mainly because participant motivation and negative psychological state often lead to premature test termination. Ameliorating the unpleasantness of this type of exercise test with the use of virtual reality technology may prolong effort expenditure during the test and result in superior performance compared to a control condition.

Additionally, improving physiological function at submaximal work rates may lead to alterations in other important testing outcomes, particularly the ventilatory threshold. The ventilatory threshold is used as a reference point for prescribing exercise intensity. An intervention that modifies this value would have repercussions for physical fitness practitioners who prescribe exercise intensity relative to the ventilatory threshold.

The general purpose of this study is to determine the effect of virtual reality on maximal aerobic exercise test performance in healthy adults. The specific questions it aims to answer are:

* Does using a virtual reality program during a maximal aerobic exercise test lead to differences in VO2peak (maximal aerobic capacity)? and,
* Does using a virtual reality program during a maximal aerobic exercise test lead to differences in work rate at the ventilatory threshold?

Secondary questions this study aims to answer include:

Does using a virtual reality program during a maximal aerobic exercise test lead to differences in

* exercise test time?
* maximal heart rate during the exercise test?
* maximal respiratory exchange ratio (RER) during the exercise test?
* heart rate (HR) at the ventilatory threshold?
* RER at the ventilatory threshold?
* psychological response [rating of perceived exertion (RPE) and affective valence] throughout the exercise test?

To address these aims, participants will complete the same maximal aerobic exercise test on a cycler ergometer under normal laboratory conditions (Control) and when viewing an immersive virtual reality video (VR). The two tests will be completed in a randomized and counterbalanced order to account for learning or familiarity effects, and will be separated by 1 week to account for the effects of testing fatigue.

Respiratory data, HR, RPE, and affective valence were collected during the exercise tests to address the aims of the study.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Answering "YES" to one or more items on the Physical Activity Readiness Questionnaire (PAR-Q).
* Women who are pregnant at the time of participation according to a pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-10-07 (Estimated); Study Completion 2024-10-07 (Estimated)

PRIMARY OUTCOMES:
VO2peak | Assessed during the exercise test for each condition.
  The highest level of oxygen uptake averaged over a 20-second period.
Ventilatory threshold | Assessed during the exercise test for each condition.
  The work load (in Watts) during the maximal cardiorespiratory exercise test at which breakpoints are identified between metabolic measures associated with the ventilatory threshold (CO2 production and O2 utilization; ventilatory equivalent for O2 and O2 utilization; and excess CO2 production).

SECONDARY OUTCOMES:
Peak power | Assessed during the exercise test for each condition.
  The work load (in Watts) of the highest exercise test stage that was completed
Total test time | Assessed during the exercise test for each condition.
  The duration of the test (in minutes), not including the warm-up.
RPE | Assessed throughout the exercise test for each condition (at the end of the warm-up and end of every even-numbered stage)..
  Rating of Perceived Exertion measured from 0 (no perceived exertion) to 10 (maximal perceived exertion).
Affective Valence | Assessed throughout the exercise test for each condition (at the end of the warm-up and end of every even-numbered stage)..
  Affective valence measured from -5 (feeling very bad) to +5 (feeling very good).
%VO2peak at ventilatory threshold | Assessed during the exercise test for each condition.
  The percentage of VO2peak at which the ventilatory threshold was reached.
Heart rate at ventilatory threshold | Assessed during the exercise test for each condition.
  The heart rate corresponding to the time that the ventilatory threshold was reached.
Heart rate at VO2peak | Assessed during the exercise test for each condition.
  The heart rate (in beats per minute) at which VO2peak was reached.
Respiratory Exchange Ratio (RER) at VO2peak | Assessed during the exercise test for each condition.
  The proportion of carbon dioxide production to oxygen consumption when VO2peak was reached.
Respiratory Exchange Ratio (RER) at ventilatory threshold | Assessed during the exercise test for each condition.
  The proportion of carbon dioxide production to oxygen consumption when the ventilatory threshold was reached.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Moore, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT06464406/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT06464406/SAP_001.pdf
  • Informed Consent Form (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT06464406/ICF_002.pdf